CLINICAL TRIAL: NCT03369535
Title: Urinary Metabolic Phenotyping of Diet-cardiovascular Disease Risk Associations: the OmniHeart Feeding Trial
Brief Title: Metabonomics to Investigate Effects of Healthy Diets on Blood Pressure: the OmniHeart Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11/LO/0773; G1002151 (Other Grant/Funding Number: MRC)
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline (Placebo Comparator): Baseline corresponds to typical American diet
  Interventions: Other: CARB rich diet; Other: MUFA rich diet; Other: PROT rich diet
- PROT rich diet (Active Comparator): Protein rich diet for 6 weeks
  Interventions: Other: CARB rich diet; Other: MUFA rich diet
- MUFA rich diet (Active Comparator): MUFA rich diet for 6 weeks
  Interventions: Other: CARB rich diet; Other: PROT rich diet
- CARB rich diet (Active Comparator): CARB rich diet for 6 weeks
  Interventions: Other: MUFA rich diet; Other: PROT rich diet

INTERVENTIONS:
Other: CARB rich diet — Consumed CARB rich diet for 6 weeks with a washout period of at least 2 weeks before the next intervention
  Arms: Baseline; MUFA rich diet; PROT rich diet
Other: MUFA rich diet — Consumed MUFA rich diet for 6 weeks with a washout period of at least 2 weeks before the next intervention
  Arms: Baseline; CARB rich diet; PROT rich diet
Other: PROT rich diet — Consumed PROT rich diet for 6 weeks with a washout period of at least 2 weeks before the next intervention
  Arms: Baseline; CARB rich diet; MUFA rich diet

SUMMARY:
To compare the urinary metabolomes on individuals undergone three different healthy diets--a carbohydrate-rich diet, a protein-rich diet, or a diet rich in unsaturated fat.

DETAILED DESCRIPTION:
BACKGROUND:

This study based on the OmniHeart dietary intervention study, a randomized, three period cross-over feeding study that compared the effects on blood pressure and plasma lipids of three DASH-like diets: a carbohydrate-rich (CARB) diet pattern, a rich in protein (PROT) and a rich in unsaturated (MUFA) fat, predominantly monounsaturated fat diet (see full details of OmniHeart dietary intervention https://clinicaltrials.gov/ct2/show/record/NCT00051350).

This metabonomic study aims to evaluate the feasibility of identifying individuals showing variation in clinical response to three different healthy diets, with the purpose of reducing cardiovascular disease (CVD) risk, using proton nuclear magnetic resonance (NMR) based metabolic phenotyping approach.

ELIGIBILITY:
Inclusion Criteria:

* with pre-hypertension (systolic BP of 120 to 139 mmHg and/or diastolic BP of 80 to 89 mmHg) or stage 1 hypertension (systolic BP of 140 to 159 mm Hg and/or diastolic BP of 90 to 99 mm Hg) and without diabetes or prior CVD

Exclusion Criteria:

* CVD or diabetes

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) | post 6 weeks intervention
  SBP reduction in mmHg

SECONDARY OUTCOMES:
Diastolic blood pressure (DBP) | post 6 weeks intervention
  DBP reduction in mmHg
low density lipoprotein cholesterol (LDL) | post 6 weeks intervention
  LDL reduction in mg/dl
high density lipoprotein cholesterol (HDL) | post 6 weeks intervention
  HDL reduction in mg/dl
triglycerides (TG) | post 6 weeks intervention
  TG reduction in mg/dl
total cholesterol | post 6 weeks intervention
  reduction in mg/dl

REFERENCES:
- [Derived] Loo RL, Zou X, Appel LJ, Nicholson JK, Holmes E. Characterization of metabolic responses to healthy diets and association with blood pressure: application to the Optimal Macronutrient Intake Trial for Heart Health (OmniHeart), a randomized controlled study. Am J Clin Nutr. 2018 Mar 1;107(3):323-334. doi: 10.1093/ajcn/nqx072. PMID 29506183